CLINICAL TRIAL: NCT05756374
Title: OUT to IN: an Outdoor Body-oriented Intervention Program to Improve Preschoolers' Social-emotional Competence
Brief Title: OUT to IN: an Outdoor Body-oriented Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Guida Veiga, Professor, University of Évora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #20088
Record Dates: First submitted 2023-02-10; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Children With Typical Development
Keywords: social-emotional development; mental health; preschool; preventive care; body-oriented interventions; play; relaxation
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OUT to IN Group (Experimental): This group will participate in biweekly sessions of psychomotricity for 10 weeks. Sessions will be implemented in the outdoors of the preschool, by a psychomotor therapist and children's teacher. Sessions will involve physical play, relaxation and expressive activities.
  Interventions: Behavioral: OUT to IN
- Control group (No Intervention): This will will maintain their usual routine at preschool.

INTERVENTIONS:
Behavioral: OUT to IN — OUT to IN comprises 20 body-oriented biweekly 40-minute sessions facilitated by a psychomotor therapist in a pedagogical partnership with the preschool teacher. Sessions are implemented outdoors. All sessions are framed in a context of freedom and self and mutual bodily resonance, according to the following structure: First, children are invited to engage in exercise play activities. Second, children engage in ludic relaxation proposals. Finally, children are asked to reflect on their bodily experiences and express themselves through different expressive mediators. Preschool teachers also participate in a 25-hour training focused on the underlying principles of OUT to In and participate in 20 body-oriented biweekly 20-minute relaxation sessions, facilitated by a psychomotor therapist.
  Arms: OUT to IN Group

SUMMARY:
The goal of this randomized trial is to examine the effects of a body-oriented intervention program on preschoolers' social-emotional competence.

The main question it aims to answer are: does OUT to IN effectively promotes preschoolers' self-awareness, self-regulation, relationship skills and motor competence? Participants are children between 3 and 6 years from portuguese preschools. The inclusion criteria are (a) participants' age between 3 and 6 years, (b) do not have participated in a similar intervention program within the last 6 months, and (c) do not have a physical condition that can affect the participation in the program. Children will be randomly allocated to the experimental group (who will participate in a 10-week intervention program with biweekly sessions of psychomotricity implemented outdoors) and to the control group (who will maintain their usual routines).

DETAILED DESCRIPTION:
Main aim: Examine the effects of a body-mind intervention program developed in outer space on motor competence and socio-emotional competence (emotional awareness, self-regulation, relationship skills) of preschool aged children.

Participants: Children attending pre-school education. Inclusion criteria are: a) attending regular pre-school education; b) not having limitations (e.g. physical limitations; intellectual deficits) to take the assessment tests; c) not having limitations to participate in the intervention sessions; d) not using drugs that can influence the dependent variables; f) not participating in a similar intervention program for at least 2 months. 250-300 children are expected to be enrolled in this study.

Children will be randomly allocated to the experimental group (who will participate in a 10-week intervention program with biweekly sessions of psychomotricity implemented outdoors) and to the control group (who will maintain their usual routines). Children will be tested before and after the intervention period.

Outcome measures:

Motor competence will be assessed through the Test of Gross Motor Development II.

Social-emotional competence will be assessed through the Study on Social and Emotional Skills questionnaire reported by parents and teachers. Parents will also fill in the Emotional Expression Questionnaire. Children will be individually tested through the recognition, identification and emotional understanding tests, the Heads Toes Knees and Shoulders test, the Day and Night test and the interoceptive accuracy test.

Stress biomarkers will also be analysed through salivary analysis. Saliva collections will be made, in a non-stimulated way, asking each child to rinse their mouth with water for about 10 seconds, swallow it and wait 30 seconds. From that moment on, all the saliva produced will be accumulated in the mouth and placed in a tube kept on ice at regular intervals. Participants will remain in a comfortable position and not speak during the collection period.

Statistical analysis: Mann-Whitney test will be used to study differences at baseline between the OUT to IN group and the control group, and to study differences in the 10- week changes between both groups. Wilcoxon Test will be used for intragroup comparisons.

ELIGIBILITY:
Inclusion Criteria:

. attending regular pre-school education;

Exclusion Criteria:

* having limitations (e.g. physical limitations; intellectual deficits) to take the assessment tests;
* having limitations to participate in the intervention sessions;
* using drugs that can influence the dependent variables;
* participating in a similar intervention program for at least 2 months.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 271 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Emotion Understanding | 10 weeks
  Will be assessed through three tasks developed by the Focus on Emotions Group (focusonemotions.nl): emotion discrimination (children are asked to place six cards, whereby they could choose between two categories happy versus unhappy faces, and angry versus sad faces cards), identification (children are asked to point to the facial expressions according to the emotion words instructed by the experimenter), and emotion attribution in a situational context (children are presented with eight illustrated emotion-evoking vignettes, designed to evoke happiness, anger, fear and sadness, and asked how the protagonist is feeling by pointing the facial expression and verbally identifying the emotion).
Self Regulation | 10 weeks
  Self-regulation is obtained through the the Day and Night task (DN), the Head Toes Knees and Shoulders task (HTKD) and the composite scale Externalizing Behaviors from the Strengths and Difficulties Questionnaire.
  In the DN task whenever the child sees a black card, must say "day", whenever the child sees a white card, must say "night".
  In the HTKS task whenever the child is asked to touch the feet, must touch the head and vice versa, when the child is asked to touch the shoulders, must touch the knees and vice versa.
  Externalizing behaviors is obtained through a composite scale which comprises two SDQ scales: behavior problems and hyperactivity. Caregivers are asked to rate their children's behavior in a 3-point likert scale, from 1 (not true) to 3 (certainly true).
Relationship skills | 10 weeks
  Empathy, Cooperation are Sociability are measured through the Study on Social and Emotional Skills Questionnaire (SSES), a caregivers and teacher report questionnaire. Caregivers and teachers were asked to fill in the Empathy (e.g. He/she can feel how others are feeling; He/she understands what others want), Cooperation (e.g., He/she works well with others; he/she likes to help others), and Sociability subscales (e.g., He/she has many friends; He/she makes friends easily) in a 5-point likert scale from one (completely disagree) to five (completely agree).
  Emotion communication is obtained through the Emotion Vocabulary Questionnaire, a caregiver-report which assesses whether children know and use emotion and/or mental state words, in a 2-point likert scale from 1 (no) to 2 (yes). The EVQ includes either basis emotions (e.g., happy, angry), complex emotions (e.g., jealous, disappointed), and mental state words (e.g. thinking, dreaming).
Interoceptive Accuracy | 10 weeks
  Interoceptive accuracy is measured through the Jumping Jack Paradigm (JJP). In the JJP task the child is first asked to sit in a chair looking at a calm screen for 3 minutes. Then examiner assesses his/her pulse to count the heart rate. Then the child is asked to choose one of the four circles, with different sizes that he/she believes it is equivalent to the heart rate. Then the child is asked to perform jumping jacks for 20 seconds. After the jumping jacks, the examiner measures her/his hear rate and asks the child to again choose one of the four circles that corresponds to his/her heart rate.
Motor Competence. | 10 weeks
  Motor Competence is assessed through the Test of Gross Motor Development-Second Edition (TGMD-2). Simple and playful exercises (throwing a ball, jumping, etc.) are performed to assess locomotion (running; galloping; hopping; leaping; jumping and sliding) and object control skills (striking; dribbling; catching; kicking; throwing and rolling). Each children performs every activity for two trials.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No